CLINICAL TRIAL: NCT04060134
Title: A Retrospective, Multi-Center, Open Label Study Evaluating SimpliDerm™ and Other Human Acellular Dermal Matrices in Breast Reconstruction
Brief Title: A Retrospective Breast Reconstruction Study
Status: Completed | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-0004
Record Dates: First submitted 2019-08-12; First posted 2019-08-16 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- SimpliDerm HADM: Patients who had SimpliDerm human acellular dermal matrix used in their breast reconstruction procedure.
  Interventions: Other: SimpliDerm HADM
- AlloDerm HADM: Patients who had AlloDerm human acellular dermal matrix used in their breast reconstruction procedure.
  Interventions: Other: AlloDerm HADM
- AlloMax HADM: Patients who had AlloMax human acellular dermal matrix used in their breast reconstruction procedure.
  Interventions: Other: AlloMax HADM
- FlexHD HADM: Patients who had FlexHD human acellular dermal matrix used in their breast reconstruction procedure.
  Interventions: Other: FlexHD HADM
- DermACELL HADM: Patients who had DermACELL human acellular dermal matrix used in their breast reconstruction procedure.
  Interventions: Other: DermACELL HADM

INTERVENTIONS:
Other: SimpliDerm HADM — Human acellular dermal matrices are used for the repair or replacement of damaged or inadequate integumental tissue or for other homologous uses of human integument.
  Groups: SimpliDerm HADM
Other: AlloDerm HADM — Human acellular dermal matrices are used for the repair or replacement of damaged or inadequate integumental tissue or for other homologous uses of human integument.
  Groups: AlloDerm HADM
Other: AlloMax HADM — Human acellular dermal matrices are used for the repair or replacement of damaged or inadequate integumental tissue or for other homologous uses of human integument.
  Groups: AlloMax HADM
Other: FlexHD HADM — Human acellular dermal matrices are used for the repair or replacement of damaged or inadequate integumental tissue or for other homologous uses of human integument.
  Groups: FlexHD HADM
Other: DermACELL HADM — Human acellular dermal matrices are used for the repair or replacement of damaged or inadequate integumental tissue or for other homologous uses of human integument.
  Groups: DermACELL HADM

SUMMARY:
To collect data on patients who have previously undergone breast reconstruction utilizing SimpliDerm and other HADMs.

DETAILED DESCRIPTION:
This study is a retrospective, multi-center, open label study evaluating SimpliDerm and other human acellular dermal matrices in breast reconstruction.

A total of up to 300 patients who underwent direct to implant (one stage) or two-stage unilateral or bilateral breast reconstruction with SimpliDerm an other HADMs at the time of implant or TE placement.

Data will be collected for a minimum of one post-surgical visit after direct implant or exchange. If more visits are available, data from those visits will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* Female patient who underwent immediate breast reconstruction post-mastectomy; either direct to implant or with a tissue expander followed by exchange for a saline or gel implant.
* HADMs such as: InteguPly, SimpliDerm, AlloDerm, FlexHD, DermACELL, Cortiva, or AlloMax used in the breast reconstruction.

Exclusion Criteria:

* Female patient who underwent cosmetic/aesthetic breast augmentation procedure or revision.
* Female patient who underwent delayed breast reconstruction procedure.
* Female patient who underwent revision of previous breast reconstruction procedure.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of up to 300 female patients, who had direct to implant or two-stage immediate breast reconstruction following unilateral or bilateral mastectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of Events | From date of surgery through study completion, an average of 9 months
  Occurrence of: infection, hematoma, seroma, capsular contracture, mastectomy skin flap dehiscence, mastectomy skin flap necrosis, expander/implant explantation, red breast syndrome, subsequent surgical interventions related to the breast reconstruction process

OTHER OUTCOMES:
Integration Assessment | From date of surgery through study completion, an average of 9 months
  Integration assessment for patients with two-stage reconstruction at time of exchange, if available, via surgeon's operative notes
Drain Removal | From date of surgery through study completion, an average of 9 months
  Time to drain removal and volume of fluid drained, if available
Intraoperative fill volume | From date of surgery through study completion, an average of 9 months
  Intraoperative fill volume

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Baptist Medical Center South, Montgomery, Alabama
  - Shoals Plastic Surgery, Muscle Shoals, Alabama
  - Tierney Plastic Surgery, Nashville, Tennessee
  - Ascension/Seton Institute of Reconstructive Plastic Surgery, Austin, Texas
  - DHR Health, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aziyo Biologics, Inc. — http://www.aziyo.com